CLINICAL TRIAL: NCT00613509
Title: Phase II Study of a Multi-Antigen Therapeutic Vaccine in Patients With Metastatic Melanoma
Brief Title: Study of a Multi-Antigen Therapeutic Vaccine in Patients With Metastatic Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: No safety concerns, the study was terminated due to slow enrollment. All enrolled patients were followed per protocol.
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MEL11
Record Dates: First submitted 2008-01-16; First posted 2008-02-13 (Estimated); Results first posted 2010-12-17 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Melanoma; Cancer
Keywords: Melanoma, Cancer
MeSH Terms: conditions — Melanoma; Neoplasms | interventions — Introns; Interferon alpha-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Study Group 1: ALVAC melanoma vaccine (Experimental): Participants will receive a multi-antigen of modified canarypox virus (ALVAC[2]) melanoma vaccine and granulocyte macrophage colony stimulating factor (GM-CSF) every 3 weeks, followed by 4 weeks of high-dose interferon alpha-2b 5 times per week.
  Interventions: Biological: ALVAC(2) Melanoma multi-antigen therapeutic vaccine
- Study Group 2: Interferon alpha-2b (Active Comparator): Participants on 4 weeks of high-dose interferon alpha-2b 5 times per week. Participants who showed disease progression after Cycle 1 will be permitted to cross over to Group 1 treatment.
  Interventions: Biological: Intron A, Interferon alpha -2b

INTERVENTIONS:
Biological: ALVAC(2) Melanoma multi-antigen therapeutic vaccine — 0.5 mL, 2 cycles
  Arms: Study Group 1: ALVAC melanoma vaccine
Biological: Intron A, Interferon alpha -2b — 0.5 mL, 5 times per week for 4 weeks
  Other Names: Intron-A®: IFN-α2b
  Arms: Study Group 2: Interferon alpha-2b

SUMMARY:
Primary objective:

To evaluate the clinical activity of the vaccine regimen, as indicated by progression-free survival versus the clinical activity of the reference treatment.

Secondary objectives:

Safety: To describe the safety profile in both treatment groups.

Efficacy: To determine the objective clinical responses of patients in both treatment groups: complete response and partial response.

DETAILED DESCRIPTION:
Eligible participants will be randomized to receive either a vaccine treatment consisting of a series of multi-antigen melanoma vaccine and GM-CSF injections, followed by high-dose IFN-α2b or only the high-dose IFN-α2b.

ELIGIBILITY:
Inclusion Criteria :

* A pathologically confirmed diagnosis of malignant melanoma with at least one measurable metastatic lesion with a minimum lesion size of 20 mm, based on radiological assessment (or 10 mm if assessed by spiral computed tomography [CT] scan ) as per Response Evaluation Criteria in Solid Tumors (RECIST) criteria (Stages IIIc, IVa, or IVb only, according to the American Joint Committee on Cancer (AJCC) staging system for melanoma). Cutaneous metastasis (assessed by physical examination) must be at least 10 mm. CT scan or magnetic resonance imaging (MRI) is required to rule out brain metastases.
* Patients who received prior treatment for their metastatic disease must have objective evidence of disease progression.
* Aged ≥ 18 years on the day of inclusion
* IRB-approved informed consent form signed
* Able to attend all scheduled visits and to comply with all trial procedures
* For a woman, inability to bear a child or negative serum pregnancy test
* For a woman of child-bearing potential, using an effective method of contraception or abstinence during the study and at least 4 weeks after the last study treatment
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 and a life expectancy of at least 6 months.
* Adequate hematologic, hepatic, and renal function (at pre-defined laboratory values).
* Fully recovered from surgery, if applicable.

Exclusion Criteria :

* Receipt of two or more previous therapies for metastatic melanoma.
* Receipt of chemotherapy or another therapy for metastatic melanoma within the last four weeks
* Receipt of adjuvant interferon therapy within the last six months
* Concurrent receipt of radiotherapy for the metastatic disease, unless for palliative purposes
* Participation in another clinical trial within the four weeks preceding the first trial treatment
* Planned participation in another clinical trial during the present trial period
* Known Human Immunodeficiency Virus (HIV) infection or hepatitis B (Ag HBs) or hepatitis C seropositivity
* Presence of active autoimmune disease (excluding vitiligo)
* Systemic hypersensitivity to bovine products or to any of the vaccine components, including egg products or Neomycin (used to prepare the vaccine), or history of a life-threatening reaction to granulocyte-macrophage colony stimulating factor (GM-CSF) or interferon (IFN)-α2b
* Current alcohol or drug addiction that may interfere with the ability to comply with trial procedures
* Significant co-morbid medical conditions, including pre-existing renal disease, cirrhosis, or major depression, which in the estimation of the investigator would preclude safe participation in the study or the accurate interpretation of data.
* A calculated glomerular filtration rate (GFR) <60 mL/min (based on the Cockroft-Gault formula).
* Previous receipt of a modified canarypox virus (ALVAC)-based vaccine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2008-06; Primary Completion 2010-04 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (19):
- United States (15):
  - Tucson, Arizona
  - Los Angeles, California
  - Aurora, Colorado
  - Atlanta, Georgia
  - Chicago, Illinois
  - St Louis, Missouri
  - Omaha, Nebraska
  - Lebanon, New Hampshire
  - Portland, Oregon
  - Bethlehem, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Greenville, South Carolina
  - Dallas, Texas
  - San Antonio, Texas
  - Madison, Wisconsin
- Canada (4):
  - Hamilton, Ontario
  - London, Ontario
  - Toronto, Ontario
  - Montreal, Quebec

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com
- See also: Related Info — http://www.cancervaccines.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 20 May 2008 to 31 March 2009 at 8 medical centers in the US and 3 medical centers in Canada.
Pre-assignment Details: A total of 23 participants who met the inclusion and exclusion criteria were enrolled and treated.
Groups:
- Study Group 1: ALVAC Melanoma Vaccine: Participants received vaccine treatment consisting of 3 series of multi-antigen ALVAC-based melanoma vaccine and GM-CSF injections, followed by four weeks of high-dose IFN-α2b. (Participants that did not show disease progression were allowed a second cycle of treatment)
- Study Group 2: Interferon Alpha-2b: Participants on Four weeks of high-dose IFN-α2b. (Participants that showed disease progression after Cycle 1 were permitted to cross over to Group 1 treatment)
Period: Cycle 1
Arm/Group | Study Group 1: ALVAC Melanoma Vaccine | Study Group 2: Interferon Alpha-2b
Started | 11 | 12
Completed | 6 (Completion of Cycle 1. 9 participants were deemed evaluable) | 4 (Completion of Cycle 1. 12 participants were deemed evaluable)
Not Completed | 5 | 8
Not completed — Adverse Event | 2 | 1
Not completed — Disease Progression | 2 | 6
Not completed — Unacceptable Toxicity | 1 | 0
Not completed — Other administrative reason | 0 | 1
Period: Cycle 2 (Group 2 = Crossover)
Arm/Group | Study Group 1: ALVAC Melanoma Vaccine | Study Group 2: Interferon Alpha-2b
Started | 11 | 4
Completed | 11 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Study Group 1: ALVAC Melanoma Vaccine | Study Group 2: Interferon Alpha-2b | Total
Number analyzed (Participants) | 11 | 12 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 10 | 19
  >=65 years | 2 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.6 (14.23) | 52.9 (14.34) | 52.8 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 5 | 7 | 12
Region of Enrollment [Number; unit: participants]
  United States | 9 | 10 | 19
  Canada | 2 | 2 | 4

OUTCOME MEASURES:

1. Other Pre Specified Outcome: Number of Participants With a Vaccine-Induced Increase of CD8 T-Cell Positive Response by Antigen
Description: The vaccine-induced increase of CD8 T-Cell positive response by antigen post-vaccination during the observation period compared to the screening values.
Time Frame: Day 0 to 32 weeks post 1st vaccination
Population: Immunologic responses were assessed in the Per-protocol evaluable population.
Measure: Number; unit: Participants
Arm/Group | Study Group 1: ALVAC Melanoma Vaccine | Study Group 2: Interferon Alpha-2b
Number analyzed (Participants) | 9 | 12
Participants
  Screening: gp100 pool1 | 0 | 0
  Screening: gp100 pool2 | 0 | 0
  Screening: gp100 pool3 | 0 | 0
  Screening: gp100 pool4 | 0 | 0
  Screening: gp100 pool5 | 0 | 0
  Screening: gp100 pool6 | 0 | 0
  Screening: NYESO-1 pool 1 | 0 | 0
  Screening: NYESO-1 pool 2 | 0 | 0
  Screening: Mart1 pool | 0 | 0
  Screening: Native 15mer pool | 0 | 0
  Screening: 9mer pool | 0 | 0
  7 Weeks post 1st Vaccination: gp100 pool1 | 0 | 0
  7 Weeks post 1st Vaccination: gp100 pool2 | 0 | 0
  7 Weeks post 1st Vaccination: gp100 pool3 | 0 | 0
  7 Weeks post 1st Vaccination: gp100 pool4 | 0 | 0
  7 Weeks post 1st Vaccination: gp100 pool5 | 1 | 0
  7 Weeks post 1st Vaccination: gp100 pool6 | 0 | 0
  7 Weeks post 1st Vaccination: NYESO-1 pool 1 | 0 | 0
  7 Weeks post 1st Vaccination: NYESO-1 pool 2 | 0 | 0
  7 Weeks post 1st Vaccination: Mart1 pool | 0 | 0
  7 Weeks post 1st Vaccination: Native 15mer pool | 0 | 0
  7 Weeks post 1st Vaccination: 9mer pool | 0 | 0

2. Other Pre Specified Outcome: Number of Participants With a Vaccine-Induced Increase of CD4 T-Cell Positive Response by Antigen
Description: The Vaccine-induced increase of CD4 T-Cell positive response by antigen post-vaccination during the observation period compared to the screening values.
Time Frame: Day 0 to 32 weeks post 1st vaccination
Population: Immunologic responses were assessed in the Per-protocol evaluable population.
Measure: Number; unit: Participants
Arm/Group | Study Group 1: ALVAC Melanoma Vaccine | Study Group 2: Interferon Alpha-2b
Number analyzed (Participants) | 9 | 12
Participants
  Screening: gp100 pool1 | 0 | 0
  Screening: gp100 pool2 | 0 | 0
  Screening: gp100 pool3 | 0 | 0
  Screening: gp100 pool4 | 0 | 0
  Screening: gp100 pool5 | 0 | 0
  Screening: gp100 pool6 | 0 | 0
  Screening: NYESO-1 pool 1 | 0 | 0
  Screening: NYESO-1 pool 2 | 0 | 0
  Screening: Mart1 pool | 0 | 0
  Screening: Native 15mer pool | 0 | 0
  Screening: 9mer pool | 0 | 0
  7 Weeks post 1st Vaccination: gp100 pool1 | 0 | 1
  7 Weeks post 1st Vaccination: gp100 pool2 | 0 | 0
  7 Weeks post 1st Vaccination: gp100 pool3 | 0 | 0
  7 Weeks post 1st Vaccination: gp100 pool4 | 0 | 0
  7 Weeks post 1st Vaccination: gp100 pool5 | 1 | 0
  7 Weeks post 1st Vaccination: gp100 pool6 | 0 | 0
  7 Weeks post 1st Vaccination: NYESO-1 pool 1 | 0 | 0
  7 Weeks post 1st Vaccination: NYESO-1 pool 2 | 0 | 0
  7 Weeks post 1st Vaccination: Mart1 pool | 0 | 0
  7 Weeks post 1st Vaccination: Native 15mer pool | 0 | 0
  7 Weeks post 1st Vaccination: 9mer pool | 0 | 0

3. Secondary Outcome: Best Overall Objective Response as Number of Participants Responding in the Intent-to-treat Population
Description: Objective response rate (ORR) is the sum of complete response (CR) and partial response (PR) Complete response = Disappearance of all target lesions. Partial response = At least a 30% decrease in the sum of longest diameter of target lesions, taking as reference the baseline sum longest diameter.
Time Frame: Day 0 to 32 weeks post 1st vaccination or treatment
Population: The best overall objective response as number of participants responding was assessed in the intent-to-treat (ITT) evaluable population.
Measure: Number; unit: Particpants
Arm/Group | Study Group 1: ALVAC Melanoma Vaccine | Study Group 2: Interferon Alpha-2b
Number analyzed (Participants) | 11 | 12
Particpants
  Participants with measurable disease at baseline | 11 | 11
  Complete Response (CR) | 0 | 0
  Partial Response (PR) | 2 | 1
  Stable Disease (SD) | 3 | 3
  Not Evaluable (NE) | 0 | 1
  Progression (PD) | 6 | 6

4. Secondary Outcome: Best Overall Objective Response in the Intent-to-treat Population
Description: as for outcome 3
Time Frame: Day 0 to 32 weeks post 1st vaccination or treatment
Population: The best overall objective response were assessed in the intent-to-treat (ITT) evaluable population.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Group 1: ALVAC Melanoma Vaccine | Study Group 2: Interferon Alpha-2b
Number analyzed (Participants) | 11 | 12
Percentage of participants | 18.2 | 9.1

5. Primary Outcome: Summary of Disease Progression in Study Participants, Intent-to-treat Population
Description: Number of evaluable study participants who had died or experienced objective disease progression (no clinical objective response to treatment as evaluated by computed tomography [CT] scans or physical examination).
Time Frame: Day 0 up to 35 weeks post 1st vaccination or treatment
Population: The Progression-Free Survival Time were assessed in the intend-to-treat (ITT) evaluable population.
Measure: Number; unit: Participants
Arm/Group | Study Group 1: ALVAC Melanoma Vaccine | Study Group 2: Interferon Alpha-2b
Number analyzed (Participants) | 11 | 12
Participants
  Progressed or died due to any cause | 7 | 6
  Did not progress or die due to any cause | 4 | 6

6. Other Pre Specified Outcome: Summary of Cellular Immune Response to the Vaccination or Treatment (Percent Regulatory T-Cells Responses)
Description: The immunogenicity of the treatment regimens was assessed by regulatory T-cell responses as assessed primarily by the multi-parametric intracellular cytokine staining (ICS) assay.
Time Frame: Day 0 to 32 weeks post 1st vaccination or treatment
Population: Immunologic responses were assessed in the per-protocol evaluable population.
Measure: Mean (Standard Deviation); unit: Percent Cell Count
Arm/Group | Study Group 1: ALVAC Melanoma Vaccine | Study Group 2: Interferon Alpha-2b
Number analyzed (Participants) | 9 | 12
Percent Cell Count
  Screening | 2.7 (1.02) | 3.4 (1.24)
  Cycle 1 Week 1 | 3.3 (1.42) | 2.3 (0.65)
  Cycle 1 Week 7 | 2.9 (0.83) | 3.1 (1.13)
  Cycle 2 Week 23 | 3.3 (0.90) | 3.8 (0.51)
  Cycle 2 Week 32 | 4.0 (0.48) | 2.6 (0.07)

7. Primary Outcome: Progression-Free Survival Time by Response Evaluation Criteria in Solid Tumor (RECIST) Criteria in the Intent-to-treat Population
Description: Progression-Free Survival was assessed by the Response Evaluation Criteria in Solid Tumor criteria from the computed tomography (CT) scans, as per-protocol
Time Frame: Day 0 - up to 35 weeks post 1st vaccination or treatment
Population: The Progression-Free Survival Time were assessed in the intend-to-treat (ITT) evaluable population.
Measure: Median (Inter-Quartile Range); unit: Weeks
Arm/Group | Study Group 1: ALVAC Melanoma Vaccine | Study Group 2: Interferon Alpha-2b
Number analyzed (Participants) | 11 | 12
Weeks | 15.9 [8.0 to NA] — NA: Upper limit not estimated because of insufficient observations above the median | 8.9 [8.3 to NA] — NA: Upper limit not estimated because of insufficient observations above the median
Statistical Analysis 1: Comparison: Study Group 1: ALVAC Melanoma Vaccine vs Study Group 2: Interferon Alpha-2b; Test type: Superiority or Other; p = 0.9406, Log Rank
Statistical Analysis 2: Comparison: Study Group 1: ALVAC Melanoma Vaccine vs Study Group 2: Interferon Alpha-2b; Test type: Superiority or Other; p = 0.9179, Likelihood ratio test

8. Secondary Outcome: Best Overall Objective Response as Mean Duration of Response (Weeks) in the Intent-to-treat Population
Description: as for outcome 3
Time Frame: Day 0 to 32 weeks post 1st vaccination or treatment
Population: The best overall objective response as mean duration of response were assessed in the intent-to-treat (ITT) evaluable population.
Measure: Mean (Full Range); unit: Weeks
Arm/Group | Study Group 1: ALVAC Melanoma Vaccine | Study Group 2: Interferon Alpha-2b
Number analyzed (Participants) | 11 | 12
Weeks | 16.3 [6.4 to 26.1] | 18.3 [18.3 to 18.3]

9. Secondary Outcome: Number of Participants Reporting a Grade 3 or Grade 4 Adverse Events by Preferred Term
Description: Common Terminology Criteria for Adverse Events (CTCAE) definitions:
  Grade 3 is a severe adverse event; Grade 4 is a life-threatening or disabling adverse event.
Time Frame: Day 0 to 12 months post last vaccination
Population: Safety assessments were conducted in the As-treated safety population.
Measure: Number; unit: Participants
Arm/Group | Study Group 1: ALVAC Melanoma Vaccine | Study Group 2: Interferon Alpha-2b
Number analyzed (Participants) | 11 | 12
Participants
  Anemia | 0 | 1
  Leukocytosis | 1 | 0
  Abdominal Pain Upper | 1 | 0
  Axillary Pain | 1 | 0
  Chest Discomfort | 1 | 0
  Chest Pain | 1 | 0
  Inflammation | 1 | 0
  Pyrexia | 0 | 1
  Sepsis | 1 | 0
  Septic Shock | 0 | 1
  Staphylococcal Bacteremia | 0 | 1
  Alanine Aminotransferase (ALT) Increased | 0 | 3
  Aspartate Aminotransferase (AST) Increased | 0 | 1
  Gamma-Glutamyl Transferase (GGT) Increased | 1 | 1
  Neutrophil Count Decreased | 1 | 0
  White Blood Cell Count Decreased | 1 | 0
  Hypernatremia | 1 | 0
  Hypoalbuminemia | 0 | 1
  Hypocalcemia | 0 | 1
  Hyponatremia | 0 | 1
  Joint Range of Motion Decreased | 1 | 0
  Metastatic Malignant Melanoma | 0 | 1
  Brain Edema | 1 | 0
  Cerebral Hemorrhage | 1 | 0
  Encephalopathy | 1 | 0
  Headache | 1 | 0
  Hemiplegia | 1 | 0
  Paraesthesia | 0 | 1
  Peripheral Sensory Neuropathy | 0 | 1
  Syncope Vasovagal | 0 | 1
  Polyuria | 1 | 0
  Hypotension | 1 | 0

ADVERSE EVENTS:
Time Frame: Adverse events data were collected from the day of vaccination for 12 months post-vaccination
Description: Due to the very limited data on the cross over participants in Group 2, Cycle 2 (n=4), cross over data were only reflected in the serious adverse event (SAE) data. Three of the 4 participants reported Gastrointestinal perforation, chest pain, disease progression, and pneumonia SAEs during the 12 months follow-up period.
Arm/Group | Study Group 1: ALVAC Melanoma Vaccine | Study Group 2: Interferon Alpha-2b
Serious Adverse Events (participants affected / at risk) | 5/11 | 5/12
Other Adverse Events (participants affected / at risk) | 5/11 | 7/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Group 1: ALVAC Melanoma Vaccine (N=11) | Study Group 2: Interferon Alpha-2b (N=12)
Gastrointestinal Perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Disease Progression (General disorders) | 2 (2) | 2 (2)
Chest Pain (General disorders) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Septic Shock (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Metastatic Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Group 1: ALVAC Melanoma Vaccine (N=11) | Study Group 2: Interferon Alpha-2b (N=12)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (2) | 0 (0)
Axillary Pain (General disorders) | 1 (2) | 0 (0)
Chest Discomfort (General disorders) | 1 (1) | 0 (0)
Inflammation (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
ALT Increased (Investigations) | 0 (0) | 3 (3)
AST Increased (Investigations) | 0 (0) | 1 (1)
GGT Increased (Investigations) | 1 (1) | 1 (1)
Neutrophil Count Decreased (Investigations) | 1 (3) | 0 (0)
White Blood Cell Count Decreased (Investigations) | 1 (3) | 0 (0)
Staphylococcal Bacteremia (Infections and infestations) | 0 (0) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Joint Range of Motion Decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Brain Edema (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral Hemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hemiplegia (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Syncope Vasovagal (Nervous system disorders) | 0 (0) | 1 (1)
Polyuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications